CLINICAL TRIAL: NCT02483286
Title: Osteoporosis and Fall Prevention With Multiple Interventions in the Metropolitan Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: The Taiwanese Osteoporosis Association. (Unknown); Wang Jhan-Yang Charitable Trust Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201503038RINB
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-01

CONDITIONS: Osteoporosis Fracture
Keywords: Osteoporosis; Fall; Fracture; sarcopenia; Exercise
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis; Fractures, Bone; Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICG (Experimental): Integrated Care Group
  Interventions: Behavioral: ICG
- MTG (Experimental): Muscle Training Group
  Interventions: Behavioral: MTG
- XBG (Experimental): X-box Group
  Interventions: Behavioral: XBG

INTERVENTIONS:
Behavioral: ICG — Core 2-hour education course including practice of study home exercise program. Weekly professional led exercise program for 90 mins at NTUHBB site with reinforcement on osteoporosis related educations and care managements from study educational booklet and CD-rom for 3-month.
  The exercise program included 15 minutes warm up with 10 minute brisk walks followed by gentle stretching. Resistance training (20-30 minutes) was provided with rubber band and bottled water (0.6-1L) as weight for major muscles of upper and lower limbs. Balance training were also provided for 10 minutes with tandem gaits and one leg standing, step up and down stairs, toe walking and heel walking.
  Subjects are encouraged to practice study home exercise program at least twice weekly.
  Arms: ICG
Behavioral: MTG — MTG group subjects were invited to NTUHBB site to receive 2 sessions of 45-minute training using isotonic strength training machines on major muscle groups each week. The intensity is set at 60-80% of 1 repetition maximum (RM). Evaluation of the exercise protocol are repeated every 2 weeks for individualized adjustments by trained physical therapist
  Arms: MTG
Behavioral: XBG — XBG group subjects were invited to LCGMH site to receive 2 sessions of 45-minute training using x-box machine with combination programs selected from existing commercial programs with a exercise training specialist.
  Arms: XBG

SUMMARY:
OBJECTIVES To determine the effects of 3 exercise interventions on sarcopenic indices among community-dwelling older adults with high osteoporotic fracture risks.

MATERIAL AND METHOD The current study enrolled subjects who screened high risk of fall, osteoporosis/fracture by standardized questionnaires or FRAX. Subjects at the National Taiwan University Hospital Bei-Hu Branch (NTUHBB) were randomized into integrated care group (ICG, target n=50) and muscle training group (MTG, target n=50). Subjects from Lingko Chang Gung Memorial Hospital (LCGMH) were all assigned into X-box group (XBG, target n=30). All participants received a CD-ROM and a one education on osteoporosis, sarcopenia, frailty, fall prevention, nutrition, and coping strategy and another hour of professional led exercise program. ICG subjects received once weekly group exercise while MTG subjects received twice weekly machine-based resistence training on major muscle groups. XBG subjects rececived twice weekly exercise with X-box based programs. Major outcomes were muscle mass (measured by bio-impedance analysis), grip strength, walking speed, and lower leg extension power at baseline and after 12-weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. older than 50 years of age
2. high risk as defined from one of the following criteria:

   * score>=1 on one minute osteoporosis risk questionnaire
   * 10 year predicted fracture risk >=20% for major osteoporotic fracture or >=3% for hip fracture from FRAX
   * fall>=2 times in pass 1 year
3. having a bone mineral density test within one year period
4. having the capability to understand the study and complete the study interventions
5. willing to participate for the intervention and study follow ups

Exclusion Criteria:

1. People younger than 50 years of age
2. Could not communicate because of hearing, visual, or cognitive problems
3. Unable to stand and walk unaided (walking aids are acceptable)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Lower extremity extensor power | 12 weeks
  Lower extremity extensor power is measured by isokinetic resistance equipment by a trained research assistant with standardized protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan